CLINICAL TRIAL: NCT07347990
Title: A Prospective, Multicenter, Single-Arm Study: Safety and Efficacy of Iptacopan in the Treatment of High-Risk Hematopoietic Stem Cell Transplantation-Associated Thrombotic Microangiopathy (TA-TMA)
Brief Title: Safety and Efficacy of Iptacopan in Patients With High-Risk Transplantation-Associated Thrombotic Microangiopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Ruijin Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Tongji Hospital (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); First Affiliated Hospital of Ningbo University (Network); Nanfang Hospital, Southern Medical University (Other); Peking University People's Hospital (Other); Fujian Medical University Union Hospital (Other); Hebei Yanda Ludaopei Hospital (Other)
Responsible Party: Principal Investigator, Yanmin Zhao, Vice Director, Bone Marrow Transplantation Center, the First Affiliated Hospital, School of Medicine, Zhejiang University, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPTA-TMA-001
Record Dates: First submitted 2025-12-27; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Thrombotic Microangiopathy; Hematopoietic Stem Cell Transplantation (HSCT)
Keywords: hematopoietic stem cell transplantation; transplantation-associated thrombotic microangiopathy; Iptacopan
MeSH Terms: conditions — Thrombotic Microangiopathies | interventions — iptacopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Iptacopan group (Experimental): This experimental arm includes patients diagnosed with transplantation-associated thrombotic microangiopathy (TA-TMA) who have failed first-line therapy; all participants will receive Iptacopan as second-line treatment.
  Interventions: Drug: iptacopan

INTERVENTIONS:
Drug: iptacopan — Iptacopan will be administered under the supervision of hospital staff during inpatient stays or self-managed by patients in an outpatient setting. The induction phase lasts 4 weeks at a dosage of 200 mg twice daily (BID). Starting from Day 29, patients will enter the maintenance phase at a dosage of 200 mg once daily (QD), continuing until treatment completion at Week 12.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of Iptacopan as a second-line treatment for high-risk hematopoietic stem cell transplantation-associated thrombotic microangiopathy (TA-TMA). Iptacopan is a selective oral small-molecule complement factor B inhibitor. It acts by inhibiting factor B, blocking the formation of C3 convertase, reducing C3b deposition, thereby suppressing C5 convertase (C3bBbC3b) and ultimately decreasing the formation of the membrane attack complex (MAC), which is expected to mitigate endothelial damage in TA-TMA pathology. The main questions this study aims to answer are:

* Does Iptacopan improve 6-month overall survival in high-risk TA-TMA patients?
* What adverse events do participants experience while taking Iptacopan?
* Does Iptacopan provide hematological response and organ function recovery in TA-TMA patients? In this prospective, multicenter, open-label, single-arm Phase II study, all participants will receive Iptacopan treatment. The primary endpoint of this study is the 6-month overall survival rate from TA-TMA diagnosis. Secondary endpoints include safety evaluation, hematological response, and organ function recovery.

During the study, participants will:

* Receive Iptacopan treatment according to protocol
* Undergo regular assessments for safety and efficacy monitoring
* Be followed for up to 24 months post-treatment initiation

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥12 years at the time of ICF signature.
2. Previous recipient of autologous or allogeneic HSCT.
3. Persistent TA-TMA despite initial management of potential triggers (e.g., CNI/mTOR inhibitor reduction, infection or GVHD treatment), with TMA activity sustained for ≥72 hours post-intervention.
4. TA-TMA diagnosis, confirmed ≤14 days prior to or during screening by either biopsy-proven microthrombi or ≥4 of the following:

(1) LDH > ULN (2) Proteinuria (rUPCR ≥1 mg/mg) (3) Hypertension (age-adjusted) (4) New-onset thrombocytopenia (platelet decrease ≥50%, count ≤50,000/mm³, or transfusion-refractory) (5) New-onset anemia or increased transfusion need (6) Microangiopathy on blood smear (schistocytes ≥1%) or biopsy (7) Elevated terminal complement complex (C5b-9) 5. High-risk TMA features (per 2023 consensus), meeting ≥1 criterion:

1. LDH ≥2× ULN
2. Elevated sC5b-9
3. Proteinuria (rUPCR ≥1 mg/mg)
4. Multi-organ dysfunction syndrome (MODS)
5. Concurrent Grade II-IV acute GVHD
6. Active systemic infection 6. Able to receive oral medication. 7. Failure of first-line therapy (e.g., CNI/mTOR inhibitor adjustment, plasma exchange, rituximab, defibrotide), excluding prior complement inhibitors.

8. Life expectancy >8 weeks. 9. Required vaccination against encapsulated bacteria (meningococcal, pneumococcal) per local guidelines, administered ≥2 weeks prior to first dose. If vaccination is delayed, antimicrobial prophylaxis is required.

10. For subjects unable to receive meningococcal vaccines, antibiotic prophylaxis must be continued throughout treatment and for 8 months post-last dose.

11. For subjects of reproductive potential: agreement to use effective contraception and, for females, a negative pregnancy test at screening.

12. Provision of signed informed consent and compliance with study procedures.

Exclusion Criteria:

1. Known familial or acquired ADAMTS13 deficiency (activity <5%).
2. Known Shiga toxin-associated HUS (positive Shiga toxin assay or culture).
3. Positive direct Coombs test with clinically significant immune-mediated hemolysis per investigator.
4. Clinically overt disseminated intravascular coagulation (DIC) according to ISTH criteria.
5. Bone marrow/graft failure.
6. Known HIV infection (confirmed by testing within 6 months prior to screening).
7. Active meningococcal disease.
8. Septic shock requiring vasopressor support within 7 days prior to enrollment.
9. Pregnant or breastfeeding.
10. Any concurrent or prior medical condition unrelated to TA-TMA that, in the opinion of the investigator or sponsor, could increase risk or confound study outcomes (e.g., significant cardiac, pulmonary, renal, endocrine, or hepatic disease).
11. All-cause respiratory failure requiring mechanical ventilation within 72 hours prior to enrollment.
12. Acute/chronic heart failure with left ventricular ejection fraction ≤40%.
13. Prior treatment with iptacopan, eculizumab, or other complement inhibitors within 60 days before first study dose.
14. Use of any investigational agent within 30 days or 5 half-lives (whichever is longer) prior to screening.
15. Recurrent primary malignancy or post-transplant lymphoproliferative disorder (PTLD).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Six-month Overall Survival Rate Following TA-TMA Diagnosis | From the date of TA-TMA diagnosis until 6 months post-diagnosis.
  The primary endpoint is defined as the proportion of patients who remain alive at 6 months after the initial diagnosis of transplantation-associated thrombotic microangiopathy (TA-TMA). Survival status will be systematically assessed through follow-up visits, medical record review, or direct patient contact at the 6-month timepoint.

SECONDARY OUTCOMES:
TA-TMA Complete Response Rate by Week 12 (Jodele Criteria) | 12 weeks from start of treatment.
  Proportion of patients achieving complete response of TA-TMA according to Jodele criteria within 12 weeks of treatment initiation.
TA-TMA Partial Response Rate by Week 12 (Jodele Criteria) | 12 weeks from start of treatment.
  Proportion of patients achieving partial response of TA-TMA (defined as response between complete response and no response) within 12 weeks of treatment initiation.
Overall Survival (OS) | Up to 24 months from diagnosis.
  Time from TA-TMA diagnosis to death from any cause.
Non-Relapse Mortality (NRM) | Up to 24 months from diagnosis.
  Time from TA-TMA diagnosis to death not attributable to hematologic disease relapse or progression.
Cumulative Incidence of Relapse (CIR) | Up to 24 months from diagnosis.
  Time from TA-TMA diagnosis to hematologic disease relapse or progression.
Mean Hemoglobin Change from Baseline | Baseline to 12 weeks.
  Change in mean hemoglobin level (g/dL) from baseline to specified time points
Exploratory Biomarker Analysis | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks after treatment .
  Exploratory analysis of complement pathway biomarkers including C5b-9 (ng/mL) and Factor B (ng/mL) levels .
Failure-Free Survival (FFS) | Up to 12 weeks from treatment initiation.
  Time (in days) from treatment initiation to first occurrence of TA-TMA response among responders.
Incidence of Acute and Chronic GVHD | Up to 24 months from treatment initiation.
  Incidence of acute and chronic graft-versus-host disease.
Multiple Organ Dysfunction Syndrome (MODS) Involvement and Resolution | Baseline, 2 weeks, 4 weeks, 8 weeks, and 12 weeks after treatment; thereafter, every three months until study completion
  Assessment of MODS organ involvement and resolution status during treatment.
Safety and Tolerability Assessment | From treatment initiation to 30 days after last dose.
  Frequency, duration, and severity of adverse events monitored through physical examinations and laboratory assessments, including infections and secondary primary malignancies. Adverse events will be graded according to CTCAE v4.03.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, China, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Risitano AM, Kulasekararaj AG, Scheinberg P, Roth A, Han B, Maciejewski JP, Ueda Y, de Castro CM, Di Bona E, Fu R, Zhang L, Griffin M, Langemeijer SMC, Panse J, Schrezenmeier H, Barcellini W, Mauad VAQ, Schafhausen P, Tavitian S, Beggiato E, Chew LP, Gaya A, Huang WH, Jang JH, Kitawaki T, Kutlar A, Notaro R, Pullarkat V, Schubert J, Terriou L, Uchiyama M, Lee LWL, Yap ES, Frieri C, Marano L, de Fontbrune FS, Gandhi S, Trikha R, Alashkar F, Yang C, Liu H, Kelly RJ, Hochsmann B, Lawniczek T, Mahajan N, Solar-Yohay S, Kerloeguen C, Ferber P, Kumar R, Wang Z, Thorburn C, Maitra S, Li S, Verles A, Dahlke M, de Latour RP. Oral iptacopan monotherapy in paroxysmal nocturnal haemoglobinuria: final 48-week results from the open-label, randomised, phase 3 APPLY-PNH trial in anti-C5-treated patients and the open-label, single-arm, phase 3 APPOINT-PNH trial in patients previously untreated with complement inhibitors. Lancet Haematol. 2025 Jun;12(6):e414-e430. doi: 10.1016/S2352-3026(25)00081-X. PMID 40447351
- [Background] Peffault de Latour R, Roth A, Kulasekararaj AG, Han B, Scheinberg P, Maciejewski JP, Ueda Y, de Castro CM, Di Bona E, Fu R, Zhang L, Griffin M, Langemeijer SMC, Panse J, Schrezenmeier H, Barcellini W, Mauad VAQ, Schafhausen P, Tavitian S, Beggiato E, Chew LP, Gaya A, Huang WH, Jang JH, Kitawaki T, Kutlar A, Notaro R, Pullarkat V, Schubert J, Terriou L, Uchiyama M, Wong Lee Lee L, Yap ES, Sicre de Fontbrune F, Marano L, Alashkar F, Gandhi S, Trikha R, Yang C, Liu H, Kelly RJ, Hochsmann B, Kerloeguen C, Banerjee P, Levitch R, Kumar R, Wang Z, Thorburn C, Maitra S, Li S, Verles A, Dahlke M, Risitano AM. Oral Iptacopan Monotherapy in Paroxysmal Nocturnal Hemoglobinuria. N Engl J Med. 2024 Mar 14;390(11):994-1008. doi: 10.1056/NEJMoa2308695. PMID 38477987
- [Background] Ardissino G, Capone V, Tedeschi S, Porcaro L, Cugno M. Complement System as a New Target for Hematopoietic Stem Cell Transplantation-Related Thrombotic Microangiopathy. Pharmaceuticals (Basel). 2022 Jul 9;15(7):845. doi: 10.3390/ph15070845. PMID 35890144
- [Background] Sartain S, Shubert S, Wu MF, Wang T, Martinez C. The alternative complement pathway activation product Ba as a marker for transplant-associated thrombotic microangiopathy. Pediatr Blood Cancer. 2020 Mar;67(3):e28070. doi: 10.1002/pbc.28070. Epub 2019 Nov 27. PMID 31774252
- [Background] Okamura H, Nakamae H, Shindo T, Ohtani K, Hidaka Y, Ohtsuka Y, Makuuchi Y, Kuno M, Takakuwa T, Harada N, Nishimoto M, Nakashima Y, Koh H, Hirose A, Nakamae M, Wakamiya N, Hino M, Inoue N. Early Elevation of Complement Factor Ba Is a Predictive Biomarker for Transplant-Associated Thrombotic Microangiopathy. Front Immunol. 2021 Jul 13;12:695037. doi: 10.3389/fimmu.2021.695037. eCollection 2021. PMID 34326846
- [Background] Jodele S, Licht C, Goebel J, Dixon BP, Zhang K, Sivakumaran TA, Davies SM, Pluthero FG, Lu L, Laskin BL. Abnormalities in the alternative pathway of complement in children with hematopoietic stem cell transplant-associated thrombotic microangiopathy. Blood. 2013 Sep 19;122(12):2003-7. doi: 10.1182/blood-2013-05-501445. Epub 2013 Jun 27. PMID 23814021
- [Background] Rotz SJ, Luebbering N, Dixon BP, Gavriilaki E, Brodsky RA, Dandoy CE, Jodele S, Davies SM. In vitro evidence of complement activation in transplantation-associated thrombotic microangiopathy. Blood Adv. 2017 Aug 23;1(20):1632-1634. doi: 10.1182/bloodadvances.2017008250. eCollection 2017 Sep 12. PMID 29296809
- [Background] Han W, Han Y, Chen J, Ma X, Chen F, Wu XJ, Qi JQ, Qiu HY, Sun AN, Wu DP. [Allogeneic hematopoietic stem cell transplantation associated thrombotic microangiopathy: 16 cases report and literature review]. Zhonghua Xue Ye Xue Za Zhi. 2016 Aug 14;37(8):666-70. doi: 10.3760/cma.j.issn.0253-2727.2016.08.007. Chinese. PMID 27587247
- [Background] Jodele S, Davies SM, Lane A, Khoury J, Dandoy C, Goebel J, Myers K, Grimley M, Bleesing J, El-Bietar J, Wallace G, Chima RS, Paff Z, Laskin BL. Diagnostic and risk criteria for HSCT-associated thrombotic microangiopathy: a study in children and young adults. Blood. 2014 Jul 24;124(4):645-53. doi: 10.1182/blood-2014-03-564997. Epub 2014 May 29. PMID 24876561
- [Background] Jodele S, Dandoy CE, Lane A, Laskin BL, Teusink-Cross A, Myers KC, Wallace G, Nelson A, Bleesing J, Chima RS, Hirsch R, Ryan TD, Benoit S, Mizuno K, Warren M, Davies SM. Complement blockade for TA-TMA: lessons learned from a large pediatric cohort treated with eculizumab. Blood. 2020 Mar 26;135(13):1049-1057. doi: 10.1182/blood.2019004218. PMID 31932840